CLINICAL TRIAL: NCT02670265
Title: Early Parenteral Nutrition in Patients With Biliopancreatic Mass Lesions (NUPAN), a Prospective Randomized Interventional Trial
Brief Title: Parenteral Nutrition in Patients With Biliopancreatic Mass Lesions
Acronym: NUPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BB61/12
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Weight Loss; Pancreatic Cancer; Biliary Tract Cancer
Keywords: malnutrition; parenteral nutrition; weight loss; pancreatic cancer; biliary tract cancer; quality of life
MeSH Terms: conditions — Weight Loss; Pancreatic Neoplasms; Biliary Tract Neoplasms; Malnutrition; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parenteral nutrition (Active Comparator): Active Comparator: Olimel peri 2.5% ® 1l/d (700 kcal/d) (Baxter GmbH, Unterschleißheim, Germany)
  Interventions: Dietary Supplement: Olimel Peri 2.5% ®
- Isotonic fluid (Placebo Comparator): Isotonic fluid 1l/d (E153, Berlin-Chemie AG, Berlin, Germany)
  Interventions: Dietary Supplement: Isotonic fluid (E153)

INTERVENTIONS:
Dietary Supplement: Olimel Peri 2.5% ® — During hospital stay patients received 1 l Olimel peri 2.5 %® containing 700 kcal (25.3 g protein, 30.0 g fat and 75.0 g glucose) daily by intravenous route.
  Arms: Parenteral nutrition
Dietary Supplement: Isotonic fluid (E153) — Controls received 1l of isotonic fluid daily by intravenous route.
  Arms: Isotonic fluid

SUMMARY:
Patients with biliopancreatic tumors are at risk for malnutrition and have to undergo many procedures for diagnostic workup that require fasting periods. In a prospective randomized monocentric study we evaluate the effect of additional parenteral nutrition on weight loss, nutritional status, quality of life and length of hospital stay.

DETAILED DESCRIPTION:
Patients with pancreatic and biliary tract cancer suffer from weight loss, malnutrition and cachexia. These factors are associated with poor prognosis, reduction in quality of life and a higher risk of complications during treatment. Moreover, patients undergo fasting periods during their diagnostic work-up at hospital that worsens malnutrition.

This is a prospective randomized monocentric study to investigate, whether parenteral nutritional supplementation may have an impact on weight loss, nutritional status, quality of life and length of hospital stay in patients with tumors of the pancreas or biliary tract. Patients either receive 1 l Olimel peri 2.5 %® (Baxter Germany GmbH Medication Delivery, Unterschleißheim, Germany containing 700 kcal, 25.3 g protein, 30.0 g fat and 75.0 g glucose) on fasting days or 1 l of isotonic fluid (E153, Berlin-Chemie AG, Berlin, Germany) in the control group. A hospital stay of at least three days is required. Patients are assessed for anthropometric measurements, bioelectrical impedance analysis, quality of life and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for suspected biliopancreatic mass lesion
* Consent to participate to the study

Exclusion Criteria:

* Liver cirrhosis (Child-Pugh B and C)
* Heart or renal failure (grade III or more)
* Dementia
* Pregnancy
* Hospital stay less than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | ≥ 3 days
  Influence of Olimel Peri 2.%% ® on body weight

SECONDARY OUTCOMES:
Nutritional status | ≥ 3 days
  Bioelectrical analysis (BIA) was performed. BCM/ECM index, phase angle, body fat were measured.
Quality of life | ≥ 3 days
  Quality of life was determined using the European EORTC QLQ-C30 form.
Length of hospital stay | ≥ 3 days
  Length of hospital stay was calculated in days.

CONTACTS AND LOCATIONS:
Overall Officials: Markus M Lerch, MD, Principal Investigator — Department of Medicine A, University Medicine Greifswald

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kruger J, Meffert PJ, Vogt LJ, Gartner S, Steveling A, Kraft M, Mayerle J, Lerch MM, Aghdassi AA. Early Parenteral Nutrition in Patients with Biliopancreatic Mass Lesions, a Prospective, Randomized Intervention Trial. PLoS One. 2016 Nov 18;11(11):e0166513. doi: 10.1371/journal.pone.0166513. eCollection 2016. PMID 27861546